CLINICAL TRIAL: NCT04566237
Title: Objective Measurements of the Opacification of the Lens After Vitrectomy
Acronym: MOCVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RLX_2020_26
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Vitrectomy; Cataract
Keywords: Objective Scatter Index (OSI); Optical Quality Analysis System (OQAS); Average Lens Density (ALD); IOLMaster® 700
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 24 months follow up after vitrectomy (Experimental): Objective Scatter Index (OSI) and Average Lens Density (ALD) at inclusion, then 3 months, 12 months and 24 months after vitrectomy
  Interventions: Procedure: Objective Scatter Index (OSI); Procedure: Average Lens Density (ALD)

INTERVENTIONS:
Procedure: Objective Scatter Index (OSI) — On Optical Quality Analysis System (OQAS) device. At Inclusion, 3 months, 12 months and 24 months after vitrectomy
Procedure: Average Lens Density (ALD) — on IOLMaster® 700 device. At Inclusion, 3 months, 12 months and 24 months after vitrectomy

SUMMARY:
Cataract is the opacification of the lens. Usually cataract occurs slowly, causing progressive vision loss over several months or years.

In ophthalmic clinical practice, repeated objective quantitative measurements of lens opacity may be necessary to document its progression and support a surgical indication.

The subjective methods of evaluating the opacification of the lens have limitations, in particular due to the lack of reproducibility between observers. Thus, innovative objective techniques with precise and reproducible cataract classification results have been developed, such as the Objective Scatter Index (OSI) on the Optical Quality Analysis System (OQAS), Visiometrics SL in 2010 and, more recently, Average Lens Density (ALD) on the IOLMaster® 700 device. Cataract is diagnosed as mature when the OSI is ≥ 2 and / or when the ALD is ≥ 74 pixel units.

Vitrectomy is a surgery of the posterior segment of the eye indicated for retinal detachment, epimacular membranes, macular holes, vitreous hemorrhage. The incidence of post-vitrectomy cataract varies among studies, and the methodology is often retrospective. Age has already been identified as a risk factor for progression since in a study of 28 eyes of patients under 50 years old, only 7% developed cataracts secondarily, compared to 79% in the 'over 50' group.

To date, there is no prospective study describing the progression kinetics of lens opacification according to precise and reproducible quantitative objective criteria in patients treated by vitrectomy. It also involves confirming the age and preoperative lens status as a risk factor for postoperative cataract progression.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old
* Indication for unilateral 3-way vitrectomy for retinal detachment, macular hole, epiretinal membrane, vitreous hemorrhage
* Bilateral phakic patient

Exclusion Criteria:

* Vitrectomy combined with cataract surgery
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Change in ALD value between baseline and 12 months after the intervention | Baseline and 12 months after vitrectomy
  ALD value : quantitative variable expressed in pixel units

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël LEJOYEUX, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (1):
- Hôpital Fondation A. de Rothschuld, Paris, France

IPD SHARING:
Plan to Share IPD: No